CLINICAL TRIAL: NCT04981457
Title: Comparative Study Between Combined Vaginal Misoprostol With Isosorbide-5-Mononitrate Versus Misoprostol Alone For Induction Of The First Trimester Missed Abortion A Randomized Clinical Trial
Brief Title: Comparative Study Between Combined Vaginal Misoprostol
Acronym: comparative
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kholod Mohamed Mahmoud Mousa Elkholy, resident of obstetrics and gynacology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-196-2021
Record Dates: First submitted 2021-07-12; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients who recieve misoprostol alone (Active Comparator): Group A (n =30 ) will receive only vaginal Misoprostol 800mcg (4 tablets Cytotec 200mcg ) ) every 3 hours to a maximum of two doses or until reaching cervical ripening or uterine contractions or bleeding assessed by the same doctor who made evaluation at the beginning.
  Interventions: Drug: Misoprostol and iso sorbide mononitrates
- patients who recieve misoprostol and iso sorbide mononitrate (Active Comparator): Group B (n =30 ) will receive combined vaginal Misoprostol 800mcg (4 tablets Cytotec ) ) every 3 hours to a maximum of two doses or until reaching cervical ripening or start of uterine contractions or bleeding. with Isosorbide-5-mononitrate (20 mg). Effox 20 mg )once at the beginning with misoprostol until reaching cervical ripening or start of and uterine contractions assessed by the same doctor who made the evaluation at the beginning.
  Interventions: Drug: Misoprostol and iso sorbide mononitrates

INTERVENTIONS:
Drug: Misoprostol and iso sorbide mononitrates — drug
  Other Names: misotac and effox

SUMMARY:
"Comparative study between Combined Vaginal Misoprostol with Isosorbide-5-Mononitrate

DETAILED DESCRIPTION:
"Comparative study between Combined Vaginal Misoprostol with Isosorbide-5-Mononitrate versus Misoprostol Alone For Induction Of The first trimester Missed Abortion A Randomized Clinical Trial"

ELIGIBILITY:
Inclusion Criteria:

* - Maternal Age 18 - 35 years.
* Gestational age first trimester of pregnancy (between 5-13 weeks).
* Missed abortion confirmed by ultrasound.
* Singleton pregnancy.
* Normal uterus and cervix on clinical examination.
* Cervix is not dilated.
* No vaginal bleeding.

Exclusion Criteria:- Evidences suggesting start of spontaneous abortion and previous trial to induce abortion.

* Presence of uterine contraction or bleeding,
* Multi-fetal pregnancy.
* Suspicion of septic abortion.
* History of Previous cervical surgery or manipulation. Ex: cervical tear , cervical cauterization .
* Uterine anomaly.
* Presence of IUD( intrauterine device) in situ
* Underlying medical diseases.Ex:diabetes mellitus,hypertension
* History of allergy or adverse effects to vaginally administered medication e.g. isosorbide -5- mononitrate
* Those unwilling to participate in the trial
* Higher order cesarean section(more than three

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Induction to abortion interval | 6 months
  Induction to abortion interval: the Duration interval between the beginning of the induction and beginning of cervical ripening assessed by cervical examination(cervix become soft and start to dilate) and uterine contractions leading to complete expulsion of the abortus spontaneous and if cervical ripening isn't occur by maximum doses the investigators will make surgical evacuation.
Number of the doses | 6 months
  the Number of the doses of misoprostol needed to complete expulsion (spontaneous or surgical)

CONTACTS AND LOCATIONS:
Overall Officials: mohamed shalaby, MD, Study Chair — Cairo u
Locations (1):
- Cairo U, Cairo, Married, Egypt

REFERENCES:
- [Background] Arteaga-Troncoso G, Villegas-Alvarado A, Belmont-Gomez A, Martinez-Herrera FJ, Villagrana-Zesati R, Guerra-Infante F. Intracervical application of the nitric oxide donor isosorbide dinitrate for induction of cervical ripening: a randomised controlled trial to determine clinical efficacy and safety prior to first trimester surgical evacuation of retained products of conception. BJOG. 2005 Dec;112(12):1615-9. doi: 10.1111/j.1471-0528.2005.00760.x. PMID 16305563
- [Background] Carlsson I, Breding K, Larsson PG. Complications related to induced abortion: a combined retrospective and longitudinal follow-up study. BMC Womens Health. 2018 Sep 25;18(1):158. doi: 10.1186/s12905-018-0645-6. PMID 30253769
- [Background] Kim C, Barnard S, Neilson JP, Hickey M, Vazquez JC, Dou L. Medical treatments for incomplete miscarriage. Cochrane Database Syst Rev. 2017 Jan 31;1(1):CD007223. doi: 10.1002/14651858.CD007223.pub4. PMID 28138973

DOCUMENTS (1):
  • Study Protocol (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT04981457/Prot_000.pdf